CLINICAL TRIAL: NCT03141294
Title: Reformative Versus Single Step Dilation Percutaneous Dilatational Tracheostomy: a Randomized Trial
Brief Title: Reformative Versus Single Step Dilation Percutaneous Dilatational Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jinhai Li, attending physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-SR-078
Record Dates: First submitted 2017-04-20; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure; Respiratory Depression
Keywords: tracheostomy，fascia，force gauge
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sd-PDT group (Placebo Comparator): The investigators applied the traditional standard dilation technique when operating tracheostomy on the standard group.
  Interventions: Procedure: reformative dilation technique
- re-PDT group (Experimental): The investigators applied the reformative dilation technique when operating tracheostomy on the re-PDT group.
  Interventions: Procedure: reformative dilation technique

INTERVENTIONS:
Procedure: reformative dilation technique — reformative dilation technique was used when operating tracheostomy
  Other Names: reformative tracheostomy

SUMMARY:
Percutaneous dilatational tracheostomy (PDT), especially single-step dilatational tracheostomy (sd-PDT), is now frequently preferred to surgical tracheostomy. Occasionally, it needs a second dilation maneuver .Dissection of the deep cervical fascia during PDT, known as reformative PDT (re-PDT), may facilitate the procedure. This study was designed to compare re-PDT with sd-PDT in ICU patients

DETAILED DESCRIPTION:
Percutaneous dilatational tracheostomy (PDT) is a popular airway management technique in the intensive care unit (ICU).Occasionally the first dilation may be challenging when using Ciaglia and colleagues' method, and a second dilation may be needed to insert the tracheostomy tube. In these circumstances, potentially life-threatening complications, such as hemorrhage and hypoxia, may arise. The investigators found the reasons for difficulty in achieving smooth dilation of the stoma.The investigators compared the traditional method with the improved method.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* requirement for long-term mechanical ventilation;
* failure of weaning from mechanical ventilation.

Exclusion Criteria:

* age <18 years;
* pre-existing infection at the tracheostomy site;
* pre-existing malignancy at the tracheostomy site;
* difficulty in identifying the anatomic landmarks;
* unstable cervical spine fracture;
* international normalized ratio (INR) >2;
* platelet count <50 000 mm3.

Ages: 44 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Force(newton) | Intraoperative (Force was measured the exact moment when investigators insert the'J' guidewire)
  Force refers to the force needed to dilate the airway and measured by force gauge

SECONDARY OUTCOMES:
Time(seconds) | Time was measured from tracheal puncture to tracheal tube placement, 180 seconds maxime
  Time refers to the time needed to finish the whole step from tracheal puncture to tracheal tube placement

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Li, Study Chair — The first Affliated Hospital with Nanjing Medical University
Locations (1):
- The Affliated Hospital wiht Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Natale G, Condino S, Stecco A, Soldani P, Belmonte MM, Gesi M. Is the cervical fascia an anatomical proteus? Surg Radiol Anat. 2015 Nov;37(9):1119-27. doi: 10.1007/s00276-015-1480-1. Epub 2015 May 7. PMID 25946970